CLINICAL TRIAL: NCT02302222
Title: The Management of Closed Surgical Incisions Resulting From Incisional Hernia Repair and/or Functional Panniculectomy Using the Prevena™ Customizable™ Dressing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHS.2012.Customizable.01
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Herniorrhaphy; Abdominoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): dry sterile dressing/gauze and steristrips
  Interventions: Device: Standard of Care Dressing
- Customizable (Experimental): Prevena Customizable Dressing with ActiV.A.C. Therapy Unit
  Interventions: Device: Customizable Dressing with ActiV.A.C. Therapy Unit

INTERVENTIONS:
Device: Customizable Dressing with ActiV.A.C. Therapy Unit
  Arms: Customizable
Device: Standard of Care Dressing
  Arms: Standard of Care

SUMMARY:
The goal of this study is to evaluate the impact of Customizable in the management of extensive closed surgical incisions for Subjects undergoing abdominal surgery for incisional hernia repair and/or functional panniculectomy as compared to SOC dressing, and to significantly reduce the SSC rate experienced by Subjects receiving Customizable vs. SOC surgical incision dressing.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

1. an adult 18 years old or older of either gender
2. able to provide their own informed consent
3. will undergo:

   1. a functional panniculectomy with a transverse or a fleur-de-lis incision

      * AND/OR -
   2. an incisional hernia repair with a vertical incision at least 20 cm in length and at least 10 cm of undermining on each side of the incision
4. BMI equal to or greater than 30
5. has maintained a stable weight for at least 3 months as determined by the Investigator (applies to post weight loss patients only)
6. pre-operatively assessed to undergo a procedure with a CDC Wound Classification of:

   1. Class I (Clean): An uninfected operative wound in which no inflammation is encountered and the respiratory, alimentary, genital or uninfected urinary tract is not entered

      * OR -
   2. Class II (Clean Contaminated): An operative wound in which the respiratory, alimentary, genital or uninfected urinary tract are entered under controlled conditions and without unusual contamination
7. willing and able to return for all scheduled study visits
8. if a female of child-bearing potential, must test negative on a urine pregnancy test
9. if a female of child-bearing potential, must be willing to utilize an acceptable method of birth control (i.e. oral contraceptives, condom with spermicide, diaphragm with spermicide, implants, IUD, injections, vaginal rings, hormonal skin patch) for the duration of the study

Intra-Operative Inclusion Criteria:

1. continues to meet all pre-operative inclusion criteria
2. has undergone a Class I or II CDC Wound Classification procedure resulting in a closed surgical incision able to be covered completely by Customizable dressing

Pre-Operative Exclusion Criteria:

1. has a systemic bacterial or fungal infection at the time of surgery for incisional hernia repair and/or functional panniculectomy
2. has a remote-site skin infection at the time of surgery for incisional hernia repair or functional panniculectomy
3. pre-operatively assessed to undergo a procedure with a CDC Wound Classification of:

   1. Class III (Contaminated): Open, fresh, accidental wounds, and/or major breaks in sterile technique or gross spillage from the gastrointestinal tract

      * OR -
   2. Class IV (Dirty-Infected): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera
4. will have a transverse or fleur-de-lis incision that extends beyond the flank area and requires moving the Subject from the supine position during surgery
5. has a known allergy or hypersensitivity to silver, or drape materials that contain acrylic adhesives
6. has participated in a clinical study within the past 30 days
7. who, in the investigator's opinion, would have any clinically significant condition that would impair the Subject's ability to comply with the study procedures

Post-Operative Exclusion Criteria:

1. found to meet any of the pre-operative exclusion criteria
2. determined to have a CDC Wound Classification of:

   1. Class III (Contaminated): Open, fresh, accidental wounds, and/or major breaks in sterile technique or gross spillage from the gastrointestinal tract

      * OR -
   2. Class IV (Dirty-Infected): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical Research Center, Miami, Florida
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Customizable: Customizable Dressing with ActiV.A.C. Therapy Unit
Period: Overall Study
Arm/Group | Standard of Care | Customizable
Started | 34 | 37
Completed | 33 | 31
Not Completed | 1 | 6
Not completed — Physician Decision | 0 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Treatment discontinued before day 5 | 0 | 1
Not completed — Withdrawn prior to any treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Standard of Care: dry sterile dressing/gauze and steristrips
  Standard of Care Dressing
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Customizable | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (7.79) | 41.8 (7.83) | 42.5 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 28 | 56
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 29 | 31 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 36 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Complications
Description: Surgical Site Complications:
  * Dehiscence
  * Surgical site infection (SSI)
Time Frame: Within 30 Days Post-Surgical Procedure
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Customizable
Number analyzed (Participants) | 34 | 35
Participants | 1 | 5
Statistical Analysis 1: Comparison: Standard of Care vs Customizable; Test type: Superiority; p = 0.1981, Fisher Exact; Risk Difference (RD) = 0.113, 95% CI 2-sided [-0.016 to 0.243]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse Events were assessed at each protocol scheduled visit. The safety population had one subject less than the ITT population as they were randomized to Standard of Care yet a received Customizable dressing. The Customizable dressing was applied without any negative pressure.
Arm/Group | Standard of Care | Customizable
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 2/36
Other Adverse Events (participants affected / at risk) | 2/34 | 7/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=34) | Customizable (N=36)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=34) | Customizable (N=36)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 5

LIMITATIONS AND CAVEATS:
The study was terminated after an interim data review as the SSC rates were outside the ranges of the sample size assumptions used for the study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT02302222/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT02302222/SAP_001.pdf